CLINICAL TRIAL: NCT00018590
Title: Center for the Study of Vascular Disease in Hispanic and Native Americans
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: MR-0087
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Vascular Disease
Keywords: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

SUMMARY:
This is a working registry of a longitudinal cohort of Hispanics, Native Americans, and non-Hispanic whites (as controls) for tracking of vascular disease endpoints. Blood samples collected for ongoing pilot projects as well as specimen banking. Pilot studies are observational and involve risk measures for stroke, atherosclerosis, and vascular inflammatory responses. Questionnaires on demographics, risk factors, and vascular disease history are performed. No interventions proposed as yet.

ELIGIBILITY:
Hispanics and Native Americans are oversampled, but non-Hispanic whites will be included for comparison purposes. No other exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2001-01

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reaven, M.D.
Locations (1):
- Southern Arizona VA Health Care System, Tucson, Arizona, United States